CLINICAL TRIAL: NCT01324999
Title: Tadalafil for Sarcoidosis Associated Pulmonary Hypertension
Acronym: SAPH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eli Lilly and Company (Industry); United Therapeutics (Industry); University of Cincinnati (Other)
Responsible Party: Principal Investigator, H. James Ford, MD, Assistant Professor of Medicine, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-2326
Record Dates: First submitted 2011-03-24; First posted 2011-03-29 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Hypertension
Keywords: Sarcoidosis Associated Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sarcoid Associated Pulm. Hypertension (Experimental): Single-arm open-label proof of concept study of tadalafil in patients with sarcoidosis associated pulmonary hypertension.
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — 20mg/day for one month then 40mg/day for additional 4 months

SUMMARY:
This study is designed to assess safety and efficacy of tadalafil in patients with Sarcoidosis Associated Pulmonary Hypertension.

Hypothesis: Tadalafil is safe and effective in treating pulmonary hypertension in patients with Sarcoidosis

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven sarcoidosis
* Mean pulmonary artery pressure > 25 mmHg at rest or greater than 30 mmHg with exercise by right heart catheterization within 1 year prior to entry into study
* Pulmonary capillary wedge pressure ≤ 15 mmHg
* PVR values ≥ 3.0 Woods units
* Forced vital capacity (FVC) > 40% predicted
* Forced expiratory volume in 1 second (FEV1) > 40% predicted
* WHO functional class II or III
* Stable sarcoidosis treatment regimen for three months prior to entry into study
* 6 minute walk distance between 150-450 meters
* Stable dose of antihypertensive medications
* On no other medication to treat PAH (sildenafil, vardenafil, treprostinil, epoprostenol, iloprost, bosentan, ambrisentan) within one month prior to enrollment and during duration of the study
* Non-pregnant females

Exclusion Criteria:

* Exercise limitation related to a non-cardiopulmonary reason (e.g. arthritis)
* Severe systemic hypertension > 170/95
* Severe systemic hypotension < 90/50
* History of priapism
* Patients with congestive heart failure (left ventricular dysfunction) LVEF < 45% by echocardiogram
* Anticipation by the investigator for escalation in sarcoidosis treatment during the course of the study
* Pulmonary hypertension related to etiology other than sarcoidosis (i.e. HIV, scleroderma, chronic thromboemboli)
* Use within 1 month of an sildenafil or vardenafil
* WHO functional class IV status
* Patients with severe other organ disease felt by investigators to impact on survival during the course of the study
* Subjects with liver function abnormalities (ALT or AST > 3 times the upper limit of normal at screening or at baseline) or chronic liver disease
* Advanced kidney failure (GFR < 30 ml/min at screening or at baseline)
* History of hypersensitivity reaction or adverse effect related to tadalafil
* Pregnant or lactating women
* Concomitant use of nitrates (any form) either regularly or intermittently
* Concomitant use of potent CYP3A inhibitors (eg, ritonavir, ketoconazole, itraconazole)
* Any additional contraindications and precautions specified in the package inserts for Tadalafil (Adcirca) not listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hubert J Ford, M.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio

REFERENCES:
- [Derived] Ford HJ, Baughman RP, Aris R, Engel P, Donohue JF. Tadalafil therapy for sarcoidosis-associated pulmonary hypertension. Pulm Circ. 2016 Dec;6(4):557-562. doi: 10.1086/688775. PMID 28090299

RESULTS

PARTICIPANT FLOW:
Groups:
- Tadalafil: 40 mg daily
Period: Overall Study
Arm/Group | Tadalafil
Started | 12
Completed | 7
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tadalafil
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 9
  White | 3
Region of Enrollment [Number; unit: participants]
  United States | 12
FEV1 [Mean (Standard Deviation); unit: percent predicted] | 58.0 (14.7)
FVC [Mean (Standard Deviation); unit: percent predicted] | 65.9 (13.4)
DLCO [Mean (Standard Deviation); unit: percent predicted] | 60.3 (25.0)
Right Atrial Pressure [Mean (Standard Deviation); unit: mm Hg] | 6.2 (4.0)
Mean Pulmonary Artery Pressure [Mean (Standard Deviation); unit: mm Hg] | 34.8 (7.1)
Pulmonary Artery Wedge Pressure [Mean (Standard Deviation); unit: mm Hg] | 10.3 (3.6)
Cardiac Index [Mean (Standard Deviation); unit: L/min/m²] | 2.4 (0.6)
Pulmonary Vascular Resistance [Mean (Standard Deviation); unit: Wood Units] | 6.2 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Distance
Time Frame: Baseline, Week 8, Week 16, Week 24
Population: Only 6 of the 7 study completers performed 6 minute walk test through week 24
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Tadalafil
Number analyzed (Participants) | 6
meters
  Baseline | 419.1 (170.1)
  Week 8 | 418.1 (143.5)
  Week 16 | 436.5 (178.1)
  Week 24 | 377.1 (140.9)
Statistical Analysis 1: Comparison: Tadalafil; Comparing baseline to week 24; Test type: Other; p = 0.68, t-test, 2 sided

2. Secondary Outcome: Resting Oxygen Saturation
Description: Percent oxygen saturation of hemoglobin as measured by pulse oximetry in the resting state.
Time Frame: Baseline, Week 24
Population: only 6 of the 7 study completers performed the 6 minute walk test through week 24.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Tadalafil
Number analyzed (Participants) | 6
percent
  Baseline | 96.5 (1.8)
  Week 24 | 95.2 (2.6)
Statistical Analysis 1: Comparison: Tadalafil; Test type: Other; p = 0.34, t-test, 2 sided

3. Secondary Outcome: Oxygen Desaturation During 6 Minute Walk Test
Description: Change (decrease) in oxygen saturation from start of 6 minute walk to nadir during the 6 minute walk test
Time Frame: Baseline, Week 24
Population: Only 6 of the 7 study completers performed the 6 minute walk test through week 24
Measure: Mean (Standard Deviation); unit: oxygen saturation percentage points
Arm/Group | Tadalafil
Number analyzed (Participants) | 6
oxygen saturation percentage points
  Baseline | 9 (6)
  Week 24 | 9 (9)
Statistical Analysis 1: Comparison: Tadalafil; Test type: Other; p = 0.99, t-test, 2 sided

4. Secondary Outcome: Maximum Borg Dyspnea Score During 6 Minute Walk Test
Description: The modified Borg scale consists of a vertical scale labelled 0 to10 with corresponding verbal expressions of progressively increasing sensation (shortness of breath) intensity. 0 represents no dyspnea, and 10 is the highest level of perceived dyspnea.
Time Frame: Baseline, Week 8, Week 16, Week 24
Population: Only 6 of the 7 study completers performed 6 minute walk test through the end of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil
Number analyzed (Participants) | 6
units on a scale
  Baseline | 4.8 (1.2)
  Week 8 | 5.0 (2.4)
  Week 16 | 5.3 (2.1)
  Week 24 | 6.3 (2.3)
Statistical Analysis 1: Comparison: Tadalafil; comparing baseline to week 24; Test type: Other; p = 0.19, t-test, 2 sided

5. Secondary Outcome: Brain Natriuretic Peptide Level
Time Frame: Baseline, Week 8, Week 16, Week 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tadalafil
Number analyzed (Participants) | 7
pg/mL
  Baseline | 58.8 (89.6)
  Week 8 | 32.3 (46.6)
  Week 16 | 37.5 (51.4)
  Week 24 | 42.6 (49.7)
Statistical Analysis 1: Comparison: Tadalafil; Comparing Baseline to week 24; Test type: Other; p = 0.68, t-test, 2 sided

6. Secondary Outcome: Short Form-36 Global Score
Description: SF- 36 investigates the standard of quality of life through a general health assessment and not specific to a particular disease, age or treatment group. It is a 36-item questionnaire measuring 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health). Each domain score ranges from 0 (worst) to 100 (best), with higher scores reflecting better health-related functional status. The global score is determined by taking an average of the individual domain scores. The global score range is from 0 (worst) to 100 (best).
Time Frame: Baseline, Week 8, Week 16, Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil
Number analyzed (Participants) | 7
units on a scale
  Baseline | 38.5 (5.3)
  Week 8 | 37.7 (6.7)
  Week 16 | 39.2 (6.5)
  Week 24 | 38.9 (8.5)
Statistical Analysis 1: Comparison: Tadalafil; comparing baseline to week 24; Test type: Other; p = 0.92, t-test, 2 sided

7. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Score
Description: The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life)
Time Frame: Baseline, Week 8, Week 16, Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil
Number analyzed (Participants) | 7
units on a scale
  Baseline | 64.5 (15.5)
  Week 8 | 65.1 (18.9)
  Week 16 | 64.3 (15.2)
  Week 24 | 71.1 (15.2)
Statistical Analysis 1: Comparison: Tadalafil; comparison of baseline to week 24; Test type: Other; p = 0.44, t-test, 2 sided

8. Secondary Outcome: Number of Participants With Change in WHO Functional Class (WHO FC)
Description: The WHO functional classification ranges from I (patient's disease does not affect daily activities) to IV (patient's disease causes severe impairment). Higher scores indicate more severe impairment.
Time Frame: Baseline, Week 24
Measure: Number; unit: participants
Arm/Group | Tadalafil
Number analyzed (Participants) | 7
participants
  Number of participants that improved to WHO FC I | 1
  Number of participants that improved to WHO FC II | 0
  Number of participants that improved to WHO FC III | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Tadalafil
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil (N=12)
Headache (Nervous system disorders) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Herpes zoster (Skin and subcutaneous tissue disorders) | 1 (1)
Influenza/pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Since this was a proof of concept study evaluating safety and tolerability of the intervention in this population, it was not powered to achieve statistical significance in changes observed from baseline to week 24 in any of the endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes